CLINICAL TRIAL: NCT01163019
Title: Utility of 2D Strain Echocardiography in Triage of Patients With Chest Pain in the Emergency Department
Brief Title: 2D Strain Echocardiography for Diagnosing Chest Pain in the Emergency Room
Acronym: 2DSPER
Status: Completed | Type: Observational
Sponsor: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Avinoam Shiran, Director, Echocardiography, Lady Davis Carmel Medical Center, Technion, Israel Institute of Technology
Other Study IDs: 2DS-CP-ED-MSS-IERG
Record Dates: First submitted 2010-07-12; First posted 2010-07-15 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Chest Pain; Coronary Artery Disease; Acute Coronary Syndrome
Keywords: Chest pain; acute coronary syndrome; Emergency department; speckle tracking imaging; 2D strain; Echocardiography
MeSH Terms: conditions — Chest Pain; Coronary Artery Disease; Acute Coronary Syndrome; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chest pain: Patients who present to the emergency department with a chief complaint of chest pain and have a moderate pre-test probability for an acute coronary syndrome

SUMMARY:
Background: Chest pain (CP) and suspected heart attack is the second most frequent complaint among patients presenting to the emergency department (ED). Present workup involves in-hospital observation for 6 - 48 hours and requires significant resources including imaging tests, some of which are invasive and involve radiation and radio-contrast agents, which can be toxic to the kidney.

CP can result from impaired blood supply to the heart muscle, which may result in impaired contraction of the heart that persists for several days. Bedside echocardiography with semi-automated speckle tracking strain analysis (2D strain) is a novel promising noninvasive tool for the evaluation of heart muscle contraction. 2D strain can be useful for evaluating patients with CP, since it can accurately detect minor impairment in heart muscle contraction that can identify patients with coronary artery disease (CAD) and impending heart attack (coronary arteries are the arteries supplying blood to the heart muscle).

Working hypothesis and aims: The investigators hypothesize that a bedside echo study with normal 2D strain may allow quick and safe ruling out of a heart attack and significant CAD disease as the cause of CP.

The main aim of the study is to validate the investigators preliminary findings in a large number of patients in order to establish whether a normal 2D strain can safely rule out a heart attack or life threatening CAD.

Methods: In a large multi-center study 1200 patients presenting to the ED with acute CP of an unclear cause will undergo echocardiography as close as possible to presentation and not more than 24 hours from cessation of pain. Patients will undergo standard workup by the ED physicians. Standard echocardiographic findings, but not the 2D strain analysis, will be made available to the attending physician. Data from discharge letters, ECGs, blood tests, stress tests, nuclear imaging, heart CT and heart catheterization will be collected. A 6-month follow-up telephone interview will be performed to collect data on survival, heart attacks, re-hospitalization and revascularization (opening heart vessels blockages). 2D strain analysis will be performed off-line in a central laboratory to evaluate the ability of 2D strain to distinguish between patients with CP from heart disease and patients without life threatening heart disease that can be early released home safely.

Expected results: The investigators expect, based on the investigators previous experience, that patients with normal 2D strain will have a very low probability of a heart attack and significant CAD. The investigators further expect these patients to have an excellent 6-month prognosis. This will allow their early and cost-effective discharge.

Importance and Probable implications to Medicine: Reduction in ED patient load and a decrease in unnecessary hospitalizations for CP. Cost and resource savings and elimination of unnecessary imaging studies, some of which are invasive or involve radiation and contrast agents.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting to the emergency department with chest pain characteristic for ischemia and suspected acute coronary syndrome and at least one of the following:

   * Planned emergency department or chest pain unit observation for at least 6 hours
   * Hospital or chest pain unit admission for suspected acute coronary syndrome
   * Planned coronary CT scan
2. Age ≥ 45 years old
3. Normal sinus rhythm
4. Patient able to give an informed consent

Exclusion Criteria:

1. ST elevation MI (≥ 1mm in at least 2 contiguous leads) or unstable patients requiring urgent care
2. Significant (≥ 1mm ST depression in at least 2 contiguous leads) on initial ECG
3. Elevated troponin on first examination
4. History of previous MI, CABG, significant Q waves on ECG or wall motion abnormality on a previous echo
5. Atrial fibrillation or abundant arrhythmia
6. CLBBB, Ventricular pacing
7. Valvular disease of at least moderate severity
8. Cardiomyopathy
9. Abnormal septal motion due to right ventricular disease or lung disease
10. Technically suboptimal echo study (> 2 segments of suboptimal quality from apical views)
11. Pregnancy
12. Inadequate strain tracing

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department with a chief complaint of chest pain
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2010-09; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Acute coronary syndrome | 1 week
Significant coronary artery disease. | 1 week

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE - death, MI or revascularization) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Avinoam Shiran, MD, Principal Investigator — Lady Davis Carmel Medical Center, Technion, Israel Institute of Technology
Locations (11):
- Israel (11):
  - Ha'Emek Medical Center,, Afula
  - Soroka University Medical Center, Beersheba
  - Hillel Yafe Medical Center, Hadera
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah-Hebrew University Medical Center, Mount Scopus, Jerusalem
  - Hadassah-University Medical Center, Ein Kerem, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Chaim Sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh Medical Center, Zrifin

REFERENCES:
- [Derived] Shiran A, Blondheim DS, Shimoni S, Jabarren M, Rosenmann D, Sagie A, Leibowitz D, Leitman M, Feinberg MS, Beeri R, Adawi S, Asmer I, Ganaeem M, Friedman Z, Liel-Cohen N. Effect of image quality on accuracy of two-dimensional strain echocardiography for diagnosing ischemic chest pain: a 2DSPER multicenter trial substudy. Int J Cardiovasc Imaging. 2019 Apr;35(4):617-625. doi: 10.1007/s10554-018-1495-x. Epub 2018 Nov 14. PMID 30430326
- [Derived] Shiran A, Blondheim DS, Shimoni S, Jabarren M, Rosenmann D, Sagie A, Leibowitz D, Leitman M, Feinberg M, Beeri R, Adawi S, Shotan A, Goland S, Bloch L, Kobal SL, Liel-Cohen N. Two-dimensional strain echocardiography for diagnosing chest pain in the emergency room: a multicentre prospective study by the Israeli echo research group. Eur Heart J Cardiovasc Imaging. 2017 Sep 1;18(9):1016-1024. doi: 10.1093/ehjci/jew168. PMID 27566720